CLINICAL TRIAL: NCT04149873
Title: Effectness of Treatment With Mechanical Insufflation-Exsufflation in Surgical Critically Ill Patients With Impaired Cough Function
Brief Title: Effectness of Treatment With Mechanical Insufflation-Exsufflation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Kuo-Chen Cheng, Principal Investigator, Chimei Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMFHR 10460(IRB10407-008)
Record Dates: First submitted 2018-01-24; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Mortality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Placebo Comparator): Control group' has the treatment with [Physical chest care ]
  Interventions: Procedure: MIE
- Experimental group-A (Placebo Comparator): 'Experimental group-A' has the treatment with [Mechanical-Insufflation- Exsufflation]
  Interventions: Procedure: MIE
- Experimental group-B (Experimental): 'Experimental group-B' has the treatment with [Mechanical-Insufflation- Exsufflation] and [Physical chest care]
  Interventions: Procedure: MIE

INTERVENTIONS:
Procedure: MIE — MIE

SUMMARY:
Patients defined with impaired cough function as maximum expiratory pressure (MEP) < 60cmH2O. Collected the patients in our surgical ICU who are able to reach 6-8CC/IBW under pressure support mode for 24 hours and MEP < 60cmH2O. Then the patients will be allocated to 3 groups to receive (1) conventional CPT (control group) (2) MI-E (study group A) (3) MI-E plus CPT (study group B) until 48 hours after extubation. Reintubation rates, ICU mortality and post-extubation ICU length of stay will be analyzed to evaluate its effects.

DETAILED DESCRIPTION:
Endotracheal intubation and mechanical ventilation are always used to treat acute respiratory failure in critically ill patients. Successful weaning from ventilator and extubation are crucial to determine the prognosis when patient's underlying disease getting improvement. The reasons for extubation failure include lack of improvement of on the work of breathing, hypoxemia, respiratory acidosis, conscious disturbance and retained respiratory secretions, etc. In our clinical practice, the factor of retained respiratory secretions plays an important role in successful extubation.

Traditional chest physiotherapy (CPT) is commonly used to help the critically patients in the effective expulsion of airway secretions. In recent years, new advanced techniques mechanical insufflations-exsufflation (MI-E) and high frequency chest wall oscillation (HFCWO)have been developed to get more effective to remove secretions for patients suffered from acute respiratory failure. The above devices have been described as an effective techniques for patients with chronic neuromuscular weakness, cystic fibrosis and bronchiectasis. By the knowledge, only one study mentioned about MI-E could reduce the reintubation rate and shorten the ICU length of stay. But its limitations include less of case number and not focusing on impaired cough function patients.

In this study, patients defined with impaired cough function as maximum expiratory pressure (MEP) < 60cmH2O. Collected the patients in our surgical ICU who are able to reach 6-8CC/IBW under pressure support mode for 24 hours and MEP < 60cmH2O. Then the patients will be allocated to 3 groups to receive (1) conventional CPT (control group) (2) MI-E (study group A) (3) MI-E plus CPT (study group B) until 48 hours after extubation. Reintubation rates, ICU mortality and post-extubation ICU length of stay will be analyzed to evaluate its effects.

ELIGIBILITY:
Inclusion criteria.

* 1.Written Informed Consent given by the patient or, if not possible, by a legally authorized representative and/or an independent physician as authorized by the competent ethics committee (EC) or independent review board (IRB) and local regulations.
* 2.To be at least 20 years of age.
* 3.To be treated in an ICU at the time of enrollment.
* 4.Endotracheal tube in place
* 5.The patient is mechanically ventilated and reach:

  1. Ventialtopr: Pressure support mode
  2. reach 6-8CC/IBW, ideal body weight for 24 hours
  3. MEP, maximum expiratory pressure < 60cmH2O

Exclusion Criteria

* 1.The patient or legally authorized representative refuse
* 2.< 20 years of age.
* 3.Neither endotracheal tube nor mechanical ventilator use
* 4.The patient is mechanically ventilated, but:

  1. The ventialtopr mode NOT: Pressure support mode
  2. No reach 6-8CC/IBW, ideal body weight for 24 hours
  3. MEP, maximum expiratory pressure > 60cmH2O
* 5.Participation as subject in another interventional study within 30 days prior to the first dose of study treatment, or planned participation in such a study during the study or within 30 days of its completion by the patient.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
mortality rate | 1 year
  One year mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chen Cheng, Chief, Study Chair — Chi Mei Medical Hospital
Locations (1):
- Department of Intensive Care Medicine; Chi Mei Medical Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No